CLINICAL TRIAL: NCT01575392
Title: Quality Assessment of Creatinines in Plasma and Urine
Brief Title: Quality Assessment Creatinines in Plasma and Urine
Status: Completed | Type: Observational
Sponsor: Medical Research Foundation, The Netherlands (Other)
Responsible Party: Principal Investigator, Nanne Kleefstra, ass. professor, Medical Research Foundation, The Netherlands
Other Study IDs: Krabbe_trial
Record Dates: First submitted 2011-11-28; First posted 2012-04-11 (Estimated); Last update posted 2012-04-11 (Estimated); Status verified 2012-04

CONDITIONS: Chronic Kidney Disease
Keywords: creatinine; chronic kidney disease; creatinine clearance; estimated glomerular filtration rate
MeSH Terms: conditions — Renal Insufficiency, Chronic

STUDY DESIGN:
Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — All patients presenting at the laboratory facility for a 24-hour creatinine clearance and patients in the dialysis population of the Isala Clinics who came for their periodical KT/V control, were informed about the study and asked to participate. From the 24-hour urine (and for peritoneal dialysis population also from the 24-hour peritoneal dialysate fluid) 4 samples of 4 ml were collected. Moreover, extra blood samples (16 ml in total) were drawn on top of the samples that were necessary for the (routine) 24-hour creatinine clearance.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patients coming for creatinine clearance: For this single group study, all patients presenting at the laboratory facility for a 24-hour creatinine clearance and patients in the dialysis population of the Isala Clinics who came for their periodical KT/V control, were informed about the study and asked to participate. Moreover, 20 'healthy' volunteers (including the investigators of this study and staff working at the clinical chemistry department of the Isala clinics) participated in this study.

SUMMARY:
In clinical practice the 24-hour creatinine clearance is often used to obtain an impression of renal function. However, the glomerular filtration rate is considered to be the best indicator of renal function. For practical and financial purposes, GFR is often estimated by means of serum creatinine based equations. These equations are also used in internation guidelines to define and classify chronic kidney disease. Therefore, accurate creatinine measurements are important to make reliable estimates of renal function. However, previous research has revealed a large variability in creatinine measurements using different measuring methods. In this study the investigators aim to establish the degree of variability in different methods to measure creatinine in a heterogenous group of Caucasian people with and without renal function loss and the influence of this variability on renal function estimating equations and the 24-hour creatinine clearance.

DETAILED DESCRIPTION:
Apart from the 24-hour creatinine clearance, also formulas to estimate the glomerular filtration rate (GFR) are increasingly used to get an impression from renal function in recent years. Based on these renal function measurements, clinical decisions are made as well as drug dose adjustments. The use of reliable serum creatinine measurements is therefore important to get accurate renal function estimates. However, serum creatinine is one of the most variable routine laboratory tests.

The importance of calibration to a traceable reference measurement of serum creatinine has been stressed. However, this standardization does not correct for analytical non-specificity problems, which occurs in certain techniques to measure creatinine, leading to under- or overestimation of the true creatinine concentration.

The aim of this cross-sectional observational study is to examine the degree of variability between diverse methods to measure creatinine in plasma and urine in a heterogenous group of Caucasian people with and without renal function loss and the influence hereof on the 24-hour creatinine clearance and the Modification of Diet in Renal Disease study equation and the consequences for chronic kidney disease staging.

ELIGIBILITY:
Inclusion Criteria:

* All patients >18 years presenting at the laboratory facility for a 24-hour creatinine clearance, or
* Persons >18 years, undergoing a renal replacing therapy by means of hemo-/peritoneal dialysis that had a KT/V appointment between May 2010 - January 2011

Exclusion Criteria:

* Patients <18 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: All patients presenting at the laboratory facility for a 24-hour creatinine clearance and patients in the dialysis population of the Isala Clinics who came for their periodical KT/V control, were informed about the study and asked to participate. Moreover, 20 'healthy' volunteers (including the investigators of this study and staff working at the clinical chemistry department of the Isala clinics) participated in this study.
Sampling Method: Probability Sample
Enrollment: 181 (Actual)
Dates: Start 2010-06; Primary Completion 2011-01 (Actual); Study Completion 2011-01 (Actual)

PRIMARY OUTCOMES:
To investigate the bias and precision between routine laboratory techniques to measure creatinine in plasma, urine and dialysate when compared to the gold standard to measure creatinine. | 6 months (plasma, urine and dialysate samples are collected only once during the running of the study)
  Creatinine concentrations of plasma, urine and/or dialysate samples will be measured using different techniques applied in daily clinical practice (jaffe, enzymatic and HPLC). For each participant creatinine will also be measured using the gold standard measure LC-MS. LCMS values will be used as reference method against which routine methods will be compared by means of absolute bias and precision per method group. Absolute bias is the mean difference between SCr values measured by individual laboratories and SCr target values; precision is defined as the SD of the absolute bias.

CONTACTS AND LOCATIONS:
Overall Officials: I Drion, MD, Principal Investigator — Diabetes Centre, Isala Clinics, Zwolle, the Netherlands; Henk JG Bilo, Prof, Study Director — Diabetes Centre, Isala Clinics, Zwolle, the Netherlands
Locations (1):
- Isala Clinics, Zwolle, Netherlands